CLINICAL TRIAL: NCT00237744
Title: CNS Plasticity Induced By Motor Learning Technologies Following Stroke
Brief Title: Brain and Coordination Changes Induced By Robotics and FES Treatment Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B3709-I
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Cerebral Stroke; Cerebrovascular Accident; Stroke
Keywords: Motor Learning; Rehabilitation; Robotics; Therapeutic Electric Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Wrist/Hand FES + Whole Arm Motor Learning (Experimental): Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning training and FES of the wrist/hand.
  Interventions: Device: Surface Functional Neuromuscular Stimulation; Other: whole arm motor learning
- Shoulder/Elbow Robotics + Whole Arm Motor Learning (Experimental): Subjects>6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning and shoulder/elbow robotics.
  Interventions: Device: Robotics training for shoulder elbow.; Other: whole arm motor learning
- Whole Arm Motor Learning (Experimental): Subjects>6 months following first stroke with diminished upper limb strength, coordination and function who received whole arm motor learning training without addition of FES or Robotics
  Interventions: Other: whole arm motor learning

INTERVENTIONS:
Device: Robotics training for shoulder elbow. — training utilizing a robot to assist with movement practice
  Arms: Shoulder/Elbow Robotics + Whole Arm Motor Learning
Device: Surface Functional Neuromuscular Stimulation — training utilizing FNS to assist with movement practice
  Arms: Wrist/Hand FES + Whole Arm Motor Learning
Other: whole arm motor learning — intervention utilizing motor learning training principles to perform part and whole task practice of meaningful everyday functional tasks.

SUMMARY:
The long-range goal of this work is to identify how to target treatment so that the brain is functionally re-organized to produce movement. This study will compare treatment response to robotics versus functional neuromuscular stimulation.

DETAILED DESCRIPTION:
Methods. Up to ninety-six chronic stroke subjects (> 12 months post stroke) will be randomized to one of the treatment groups: Wrist/hand Functional Electrical Stimulation (FES)+whole arm motor learning group; shoulder/elbow robotics + whole arm motor learning group; and whole arm motor learning group. For all groups, treatment will offered 5 hrs/day, 5 days/week, for 12 weeks. All three treatment groups will receive motor learning therapy. For the Wrist/hand FES+whole arm motor learning group, there will be the addition of FES during treatment. For the Shoulder/elbow robotics + whole arm motor learning group there will be the addition of robotics training. Outcome measures will be collected at weeks 1, 6, 12, and three months after the end of treatment. Measures will include muscle strength (Manual Muscle Testing); coordination of joint movement (Fugl-Meyer Coordination Scale); motor control of target acquisition, pathway maintenance; and smoothness of movement (robotics measures); performance of 13 functional tasks (Arm Motor Ability Test); and quality of life (Stroke Impact Scale). Measures of brain function will be non-invasive and will include cognitive planning time, cognitive effort level, and location of brain activity during simple shoulder and arm movements. Changes in brain function measures will reflect plasticity or adaptability in response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and at least 12 months post stroke.
* Difficulty using upper limb for functional tasks.
* Age >21 years

Exclusion Criteria:

uncontrolled, chronic medical condition

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, PhD MS, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Background] Fang Y, Yue GH, Hrovat K, Sahgal V, Daly JJ. Abnormal cognitive planning and movement smoothness control for a complex shoulder/elbow motor task in stroke survivors. J Neurol Sci. 2007 May 15;256(1-2):21-9. doi: 10.1016/j.jns.2007.01.078. Epub 2007 Mar 27. PMID 17391704
- [Background] Fang Y, Daly JJ, Sun J, Hvorat K, Fredrickson E, Pundik S, Sahgal V, Yue GH. Functional corticomuscular connection during reaching is weakened following stroke. Clin Neurophysiol. 2009 May;120(5):994-1002. doi: 10.1016/j.clinph.2009.02.173. Epub 2009 Apr 10. PMID 19362515
- [Background] Daly JJ, Hrovat K, Holcomb J, Pundik S. Brain control of functional reach in healthy adults and stroke survivors. Restor Neurol Neurosci. 2014;32(5):559-73. doi: 10.3233/RNN-130361. PMID 24613940
- [Background] Kisiel-Sajewicz K, Fang Y, Hrovat K, Yue GH, Siemionow V, Sun CK, Jaskolska A, Jaskolski A, Sahgal V, Daly JJ. Weakening of synergist muscle coupling during reaching movement in stroke patients. Neurorehabil Neural Repair. 2011 May;25(4):359-68. doi: 10.1177/1545968310388665. Epub 2011 Feb 22. PMID 21343527
- [Background] Wang XF, Jiang Z, Daly JJ, Yue GH. A generalized regression model for region of interest analysis of fMRI data. Neuroimage. 2012 Jan 2;59(1):502-10. doi: 10.1016/j.neuroimage.2011.07.079. Epub 2011 Jul 31. PMID 21839177
- [Background] Daly JJ, Hrovat K, Pundik S, Sunshine J, Yue G. fMRI methods for proximal upper limb joint motor testing and identification of undesired mirror movement after stroke. J Neurosci Methods. 2008 Oct 30;175(1):133-42. doi: 10.1016/j.jneumeth.2008.07.025. Epub 2008 Aug 22. PMID 18786565
- [Derived] Philips GR, Daly JJ, Principe JC. Topographical measures of functional connectivity as biomarkers for post-stroke motor recovery. J Neuroeng Rehabil. 2017 Jul 6;14(1):67. doi: 10.1186/s12984-017-0277-3. PMID 28683745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by word of mouth and from an advertisement flyer.
Groups:
- Wrist/Hand FES + Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning and wrist/hand FES.
- Shoulder/Elbow Robotics + Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning and shoulder/elbow robotics.
- Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning.
Period: Overall Study
Arm/Group | Wrist/Hand FES + Whole Arm Motor Learning | Shoulder/Elbow Robotics + Whole Arm Motor Learning | Whole Arm Motor Learning
Started | 11 | 11 | 18
Completed | 8 | 10 | 18
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Shoulder/Elbow Robotics + Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, and impairment of shoulder/elbow > wrist hand.
- Wrist/Hand FES + Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, and impairment of wrist hand >shoulder/elbow
- Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, and impairment of shoulder/elbow=wrist hand
- Total: Total of all reporting groups
Arm/Group | Shoulder/Elbow Robotics + Whole Arm Motor Learning | Wrist/Hand FES + Whole Arm Motor Learning | Whole Arm Motor Learning | Total
Number analyzed (Participants) | 11 | 11 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 13 | 31
  >=65 years | 2 | 2 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 8 | 6 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: AMAT
Description: The AMAT is a measure of complex functional task performance of a variety of specified tasks and is measured in seconds summed across the various tasks. A higher score is indicative of decreased performance on the measure. A max score of 3000 seconds would indicate inability to perform any portion of the test.
Time Frame: prior to treatment and following 3 months of treatment
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Shoulder/Elbow Robotics+Whole Arm Motor Learning: Subjects>6 months following first stroke with diminished upper limb strength, coordination and function, who received whole arm motor learning and shoulder/elbow robotics.
- Wrist/Hand FES+Whole Arm Motor Learning: The intervention provided in this group included surface FES and whole are motor learning.
- Whole Arm Motor Learning Group: Interventions included whole arm motor learning, FES and Robotics.
Arm/Group | Shoulder/Elbow Robotics+Whole Arm Motor Learning | Wrist/Hand FES+Whole Arm Motor Learning | Whole Arm Motor Learning Group
Number analyzed (Participants) | 10 | 8 | 18
seconds
  Pre Treatment AMAT | 1693 (631) | 1693 (947) | 1556 (703)
  Post Treatment AMAT | 1386 (572) | 1341 (900) | 1187 (703)

2. Primary Outcome: M1 Activation Absolute Change Score
Description: A measure of brain activation change in the area of M1 following intervention (pre to post intervention). A number greater than 0 indicates a change in brain activation in the area of M1. The maximum voxel activation for a healthy adult in the studied region of Interest (M1) is 659.
Time Frame: at baseline and following 3 months of treatment
Population: This is a sub sample of subjects eligible to undergo fMRI testing. A total of 23 subjects were eligible (5 subjects in the wrist/hand FES+ whole arm motor learning group; 8 subjects in the shoulder/elbow robotics+whole arm motor learning group and 10 subjects in the Whole arm motor learning group).
Measure: Mean (Standard Deviation); unit: voxels
Arm/Group | Wrist/Hand FES + Whole Arm Motor Learning | Shoulder/Elbow Robotics + Whole Arm Motor Learning | Whole Arm Motor Learning
Number analyzed (Participants) | 5 | 8 | 10
voxels | 359.6 (323.3) | 489.88 (505.8) | 429.7 (327.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of study participation.
Groups:
- Wrist/Hand FES + Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, and impairment of wrist/hand> shoulder/elbow.)
- Whole Arm Motor Learning: Subjects > 6 months following first stroke with diminished upper limb strength, coordination and function, and impairment of shoulder/elbow = wrist hand.
Arm/Group | Wrist/Hand FES + Whole Arm Motor Learning | Shoulder/Elbow Robotics + Whole Arm Motor Learning | Whole Arm Motor Learning
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/18
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes